CLINICAL TRIAL: NCT03499964
Title: ROBUST III - Re-Establishing Flow Via Drug Coated Balloon For The Treatment Of Urethral Stricture Disease - A Randomized Control Trial
Brief Title: ROBUST III- Re-Establishing Flow Via Drug Coated Balloon For The Treatment Of Urethral Stricture Disease
Acronym: ROBUST-III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Collaborators: Laborie Medical Technologies Inc. (Industry); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR1076
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Urethral Stricture
Keywords: pivotal trial; randomized; lower urinary tract symptoms (LUTS); urethral stricture; obstruction
MeSH Terms: conditions — Urethral Stricture; Lower Urinary Tract Symptoms; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Optilume Treatment (Experimental): The treatment arm will be the Urotronic Optilume Drug Coated Balloon (DCB).
  Interventions: Device: Optilume Drug Coated Balloon (DCB)
- Control Treatment (Active Comparator): The control arm will be treated by a urethral dilation method considered to be best standard of care for the study site and subject. A control treatment may be either a rod, uncoated balloon or DVIU.
  Interventions: Device: Control Treatment

INTERVENTIONS:
Device: Optilume Drug Coated Balloon (DCB) — The Optilume Drug Coated Balloon (DCB) is a guidewire compatible catheter with a tapered atraumatic tip. The distal end of the catheter has an inflatable balloon coated with a proprietary coating containing the drug paclitaxel that facilitates the drug's transfer to the urethral wall upon inflation.
  Arms: Optilume Treatment
Device: Control Treatment — A control subject may be dilated with either a rod, uncoated balloon or DVIU until the desired result is reached, based on standard of care for the clinical site and treating physician
  Other Names: Uncoated dilation balloon; Direct Vision Internal Urethrotomy (DVIU); Rigid Rod
  Arms: Control Treatment

SUMMARY:
ROBUST III is a prospective, multi-center, randomized controlled adaptive sample size clinical trial to establish the safety and effectiveness for the Optilume Stricture Drug Coated Balloon (DCB).

DETAILED DESCRIPTION:
ROBUST III is a prospective, multi-center, single blind randomized controlled clinical trial in a 2:1 allocation of treatment versus control device.

This study is an adaptive design with an interim analysis for sample size re-estimation performed after 60 subjects have been enrolled. The interim analysis will be be undertaken following completion of the 6-month follow-up data from these subjects. Based on the results of the interim analysis, the final total sample size required for the study will be re-estimated. A minimum of 140 subjects, and a maximum of 200 subjects (pending the re-estimation) will be enrolled in the study. A Data Monitoring Committee (DMC) will review the interim analysis results, including the sample size re-estimation and make recommendations related to trial continuation to the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years' old
2. Visual confirmation of stricture via cystoscopy or urethrogram
3. Single, tandem or diffuse anterior urethral stricture(s), less than or equal to 3.0 cm total length measured by retrograde urethrogram. (Stricture length is defined as the distance between the most distal edge of the stricture to the most proximal edge of the stricture).
4. Two or more prior dilation treatments of the same stricture, including DVIU (Direct Vision Internal Urethrotomy), but no prior urethroplasty.
5. Significant symptoms of stricture such as frequency of urination, dysuria, urgency, hematuria, slow flow, feeling of incomplete emptying, recurrent urinary tract infections (UTI's).
6. International Prostrate Symptoms Score (IPSS) score of 11 or higher (assumed to be "35" if suprapubic catheter is present)
7. Lumen diameter ≤ 12F by urethrogram
8. Qmax <15 ml/sec (assumed to be "0" if suprapubic catheter is present)
9. Guidewire must be able to cross the lesion

Exclusion Criteria:

1. Subjects with diffuse stricture length, greater than 3.0 cm in total length. (Stricture length is defined as the distance between the most distal edge of the stricture to the most proximal edge of the stricture).
2. Subjects with a history of hypersensitivity reactions to TAXOL, on medication that may have negative interaction with paclitaxel, with solid tumors who have a baseline neutrophil counts of <1500 cells/mm3 or subjects with AIDS-related Kaposi's sarcoma with baseline neutrophile counts of <1000 cells/mm3.
3. Subjects who had an indwelling suprapubic catheter longer than three (3) months total prior to enrollment.
4. Previous urethroplasty within the anterior urethra
5. Stricture dilated or incised within the last six (6) weeks (urethral catheterization is not considered dilation)
6. Presence of local adverse factors, including abnormal prostate making catheterization difficult, urethral false passage or fistula.
7. Presence of signs of obstructive voiding symptoms not directly attributable to the stricture at the discretion of the physician
8. Diagnosis of untreated and unresolved BPH or BNC
9. Untreated stress urinary incontinence (SUI).
10. History of diagnosed radiation cystitis.
11. Diagnosis of carcinoma of the urethra, bladder or prostate within the last two (2) years
12. Active kidney, bladder, urethral or ureteral stone passage in the last six (6) weeks or concern of stone passage in the next 6 weeks at the discretion of the investigator.
13. Diagnosis of chronic renal failure and treatment with hemodialysis
14. New diagnosis of OAB (overactive bladder) within the last six (6) months
15. Use of alpha blockers, beta blockers, OAB (Overactive Bladder) medication, anticonvulsants (drugs that prevent or reduce the severity and frequency of seizures), and antispasmodics where the dose is not stable. (Stable dose is defined as having the same medication and dose in the last six months.)
16. Dependence on Botox (onabotulinumtoxinA) in urinary system
17. Presence of an artificial urinary sphincter, slings, or stent(s) in the urethra or prostate
18. Known neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function
19. Diagnosed with Lichen Sclerosus, or stricture due to balanitis xerotica obliterans (BXO)
20. Previous hypospadias repair
21. History of cancer in non-genitourinary system which is not considered in complete remission (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered in complete remission if there has been no evidence of cancer within two (2) years of enrollment
22. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires
23. Unwilling to use protected sex for thirty (30) days' post treatment
24. Unwilling to abstain or use protected sex for ninety (90) days post treatment if sexual partner is of child bearing potential.
25. Inability to provide Informed Consent Form (ICF) and/or comply with all the required follow-up requirements
26. Participation in other pre-market studies or treatment with an investigational drug or device. Long term follow up or post market study of an approved device is allowed.
27. Current active infection in the urinary system
28. Current uncontrolled diabetes (hemoglobin A1c > 8.0%) or evidence of poor wound healing due to diabetes
29. Diagnosed or suspected primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function, sphincter function or poor detrusor muscle function.
30. Visible hematuria in subject's urine sample without known contributing factor
31. Invisible hematuria (or significant microscopic hematuria, i.e. hematuria of ≥ 3 RBC's/HPF) that may be caused by a clinically significant disease unless it is attributed to the urethral stricture disease or other causes which are benign and not requiring treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Elliott, MD, Principal Investigator — University of Minnesota; Ramon Virasoro, MD, Principal Investigator — US Department of Veterans Affairs
Locations (22):
- United States (21):
  - Academic Urology and Urogynecology of Arizona, Phoenix, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Advanced Urology Institute, Daytona Beach, Florida
  - University of Iowa, Iowa City, Iowa
  - Chesapeake Urology Research, Annapolis, Maryland
  - Chesapeake Urology, Hanover, Maryland
  - University of Minnesota Department of Urology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - Adult & Pediatric Urology, PC, Omaha, Nebraska
  - New Jersey Urology, Voorhees Township, New Jersey
  - Western New York Urology Associates, Cheektowaga, New York
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - Iris Cantor Men's Health Center, New York, New York
  - Integrated Medical Professionals OBP, North Hills, New York
  - Carolina Urology Partners, Concord, North Carolina
  - Oregon Urology Institute, Springfield, Oregon
  - UT Southwestern, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
- Royal Victoria Hospital, Glen Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elliott SP, Coutinho K, Robertson KJ, D'Anna R, Chevli K, Carrier S, Aube-Peterkin M, Cantrill CH, Ehlert MJ, Te AE, Dann J, DeLong JM, Brandes SB, Hagedorn JC, Levin R, Schlaifer A, DeSouza E, DiMarco D, Erickson BA, Natale R, Husmann DA, Morey A, Olsson C, Virasoro R. One-Year Results for the ROBUST III Randomized Controlled Trial Evaluating the Optilume(R) Drug-Coated Balloon for Anterior Urethral Strictures. J Urol. 2022 Apr;207(4):866-875. doi: 10.1097/JU.0000000000002346. Epub 2021 Dec 2. PMID 34854748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optilume Treatment | Control Treatment
Started | 79 | 48
Completed | 68 | 21
Not Completed | 11 | 27
Not completed — Lack of Efficacy | 6 | 26
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optilume Treatment | Control Treatment | Total
Number analyzed (Participants) | 79 | 48 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (15.5) | 60.6 (16.0) | 59.4 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 79 | 48 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 75 | 45 | 120
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 65 | 39 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 2 | 6
  United States | 75 | 46 | 121
Stricture Etiology [Count of Participants; unit: Participants]
  Iatrogenic | 21 | 16 | 37
  Idiopathic | 42 | 22 | 64
  Inflammatory | 1 | 2 | 3
  Traumatic | 14 | 7 | 21
  Unknown | 1 | 1 | 2
Anatomic Stricture Location [Count of Participants; unit: Participants]
  Bulbar Urethra | 71 | 45 | 116
  Penile Urethra | 8 | 2 | 10
  Unknown | 0 | 1 | 1
Stricture Length [Mean (Standard Deviation); unit: cm] | 1.63 (0.76) | 1.72 (0.73) | 1.67 (0.75)
Prior Dilations [Median (Standard Deviation); unit: Dilations] | 3.0 (1.73) | 3.0 (7.7) | 3.0 (4.78)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Stricture Free
Description: The percentage of subjects deemed to be stricture free will be compared between arms. Stricture free subjects are those for which a 16F flexible cystoscope or 14F Foley catheter is able to be passed through the treated stricture without significant resistance.
Time Frame: 6 months
Population: Only subjects with cystoscopy completed at 6 month visit or with known repeat intervention were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume Treatment | Control Treatment
Number analyzed (Participants) | 67 | 41
Participants | 50 | 11
Statistical Analysis 1: Comparison: Optilume Treatment vs Control Treatment; Test type: Superiority; p < 0.0001, Chi-squared, Corrected

2. Primary Outcome: Safety: Rate of Major Device or Procedure Related Complications
Description: Rate of Major Device or Procedure Related complications
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume Treatment | Control Treatment
Number analyzed (Participants) | 79 | 48
Participants | 0 | 0

3. Secondary Outcome: Change in Qmax (Peak Flow Rate)
Description: Change in peak urinary flow rate (Qmax) from baseline to 6 months post treatment. Positive values indicate an increase in Qmax from baseline to 6 months, while negative values indicate a decrease in Qmax.
Time Frame: 6 months
Population: Patients with a measured Qmax at baseline and 6 months. Subjects that underwent repeat treatment for a recurrent stricture had the last observed Qmax value prior to repeat treatment utilized (worst case imputation).
Measure: Mean (Standard Deviation); unit: mL/Sec
Arm/Group | Optilume Treatment | Control Treatment
Number analyzed (Participants) | 67 | 44
mL/Sec | 8.8 (9.2) | 4.1 (7.2)
Statistical Analysis 1: Comparison: Optilume Treatment vs Control Treatment; Test type: Superiority; p = 0.003, t-test, 2 sided

4. Secondary Outcome: IPSS Percent Responder (50% Improvement in IPSS Score)
Description: The proportion of subjects considered to be therapeutic responders, defined as an improvement of greater than or equal to 50% in the International Prostate Symptom Score [IPSS] without repeat intervention, in the Optilume DCB arm at 12 months will be compared to a performance goal of 50%. The IPSS was developed to measure symptom severity for bladder outlet obstruction, with a range of 0 (no symptoms) to 35 (worst possible symptoms).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume Treatment
Number analyzed (Participants) | 59
Participants | 39

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Adverse event collection began at the time of randomization. Subjects were queried about adverse events occuring since last contact at each study visit.
Arm/Group | Optilume Treatment | Control Treatment
All-Cause Mortality (participants affected / at risk) | 1/79 | 0/48
Serious Adverse Events (participants affected / at risk) | 9/79 | 8/48
Other Adverse Events (participants affected / at risk) | 51/79 | 38/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume Treatment (N=79) | Control Treatment (N=48)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral Cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Thalmus Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal Infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Anesthetic Complication - Pulmonary (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume Treatment (N=79) | Control Treatment (N=48)
Urethral Stenosis (Renal and urinary disorders) | 9 (9) | 20 (20)
Dysuria (Renal and urinary disorders) | 7 (7) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 6 (7) | 4 (4)
Bladder Spasm (Renal and urinary disorders) | 4 (4) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 7 (16) | 5 (8)
Bacteriuria (Infections and infestations) | 5 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Post-Procedure Hematuria (Injury, poisoning and procedural complications) | 9 (9) | 2 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03499964/Prot_SAP_000.pdf